CLINICAL TRIAL: NCT00759577
Title: Feasibility of "At-home" Titration of Solifenacin 5 and 10mg and Effect on Symptoms and Quality of Life in a Typical OAB Population
Brief Title: Feasibility of "At-home" Titration of Solifenacin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty with enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Benjamin Brucker, Clinical Instructor, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VESI-8E01
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Home titration (Other): Patients were given drug to self titrate
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — 5mg and 10 mg, oral once daily
  Other Names: Vesicare

SUMMARY:
This is an open-label single center trial to study improvements in symptom bother and quality of life in overactive bladder patients self titrating solifenacin 5mg and 10 mg. The study is designed to reflect real world conditions in typical male and female OAB patients presenting for treatment.

DETAILED DESCRIPTION:
Open-label single center trial to study improvements in symptom bother and quality of life in OAB patients self titrating solifenacin 5mg and 10 mg. The study was designed to reflect real world conditions in typical male and female OAB patients presenting for treatment. After eligibility was confirmed, subjects completed a number of questionnaires which include patient perception of bladder condition (PPBC)12, Overactive Bladder Questionaire (OAB-q13), visual analog scale (VAS) 0-100 assessing bother of urge incontinence, urgency, frequency and nocturia over the past week.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory male or female patients aged ≥18 years of age and able to use the toilet without difficulty.
2. Symptoms of OAB for > 3 months.
3. Written informed consent (IC) has been obtained.
4. Capable of filling out questionnaires.
5. Patients may be included if they were never exposed to anticholinergic agents specified for the treatment of OAB. Patients may also be included if they have previously been treated with FDA-approved anticholinergic agents for the treatment of OAB such as oxybutynin chloride (generic oxybutynin chloride, Ditropan XL®, Ditropan®, or OxytrolTM), tolterodine tartrate (Detrol® or Detrol LA®), or trospium chloride (Sanctura®, Sanctura XR®) and are no longer receiving such treatment for at least 14 days.
6. Patients undergoing non-medical treatments for OAB (pelvic floor exercises or any behavioral modification) must have had treatment initiated at least 4 weeks prior to enrollment and should not change regimen.
7. Normal urine analysis or sterile urine specimen (culture negative)

Exclusion Criteria:

1. Previous treatment with darifenacin
2. Duration of urgency with or without urge incontinence, usually accompanied with frequency and nocturia for <3 months
3. Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the Investigator
4. Evidence of a urinary tract infection (UTI); chronic inflammation such as interstitial cystitis and bladder stones
5. Clinically significant outflow obstruction (benign prostatic hyperplasia [BPH]) as determined by the Investigator.
6. Uncontrolled narrow angle glaucoma, urinary or gastric retention
7. All patients with severe renal or hepatic impairment will be excluded from the trial; dose increases to 10mg are not permitted for patients that have moderate hepatic impairment as evidenced by liver function testing.
8. Women of childbearing potential who are pregnant or intend to become pregnant during the study or who are sexually active and practicing an unreliable method of birth control, as judged by the Investigator, or will be lactating during the study.
9. A history of bladder cancer
10. Known or suspected hypersensitivity to solifenacin succinate, any of its components (lactose monohydrate, corn starch, hypromellose 2910, magnesium stearate, talc, polyethylene glycol 8000 and titanium dioxide with yellow ferric oxide [5mg tablet] or red ferric oxide [10 mg tablet]), or other anticholinergics.
11. Participation in any clinical trial (except patient registry trial) involving an investigational drug, within 30 days prior to enrollment
12. Patients with chronic severe constipation or history of diagnosed gastrointestinal disease obstruction.
13. Patients with hematuria.
14. Any clinical condition, which, in the opinion of the Investigator, would not allow safe completion of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the planned 100 patients to be enrolled only 36 were enrolled.
Groups:
- At Home Titration: Starting with 5mg of solifenacin by mouth daily with self-titration ("at home") up 10mg of solifenacin by mouth daily.
Period: Overall Study
Arm/Group | At Home Titration
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | At Home Titration
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants] — No participants were analyzed because completed questionnaires were not returned. Secondary to poor enrollment the study was terminated and efforts were not made to gather this data after termination
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline gender of those that actually started medication was not available. The study was terminated early secondary to poor enrollment. Efforts to collect this data after closure was not made.

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Patient Perception of Bladder Condition Score (PPBC)
Description: Difference in Patient Perception of Bladder Condition (PPBC) score from start of medication to end of trial (12 weeks). This is a single item patient reported global question that assesses a patients subjective impression of the current urinary problems. The patients is asked to rate their perceived bladder condition on a 6 point scale ranging from 1 (no problem) at all to 6 (many severe problems). To assess change in PPBC the baseline value is subtracted from the end of study value. Thus changes in score typically range from -2 to 2. Negative values represent an improvement.
Time Frame: 12 weeks
Population: There was no questionnaire available for analysis. Secondary to poor enrollment the study was stopped and efforts to collect questionnaires at an earlier time point were not carried out.
Arm/Group | At Home Titration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Serious adverse events were not collected/assessed at the end of study. The study was terminated secondary to poor enrollment and data on serious adverse events was not collected at time of termination (prior to 12 weeks). Other adverse events were not collected/assessed at the end of study or at the time of termination.
Arm/Group | At Home Titration
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No